CLINICAL TRIAL: NCT01758081
Title: Effects of Vitamin D and Omega-3 Fatty Acids on Infectious Diseases and hCAP18
Brief Title: Effects of Vitamin D and Omega-3 Fatty Acids on Infectious Diseases and hCAP18 (VITAL Infection)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Carlos A. Camargo, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AI093723
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Infections; Human Cathelicidin Antimicrobial Peptide (hCAP-18)
MeSH Terms: conditions — Infections | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- vitamin D + fish oil (Active Comparator): vitamin D3 + Omacor
  Interventions: Dietary Supplement: vitamin D3; Drug: omega-3 fatty acids (fish oil)
- vitamin D + fish oil placebo (Active Comparator): vitamin D3 + fish oil placebo
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: fish oil placebo
- vitamin D placebo + fish oil (Active Comparator): vitamin D placebo + Omacor
  Interventions: Drug: omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3 placebo
- vitamin D placebo + fish oil placebo (Placebo Comparator): vitamin D placebo + fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: fish oil placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day
  Arms: vitamin D + fish oil; vitamin D + fish oil placebo
Drug: omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Arms: vitamin D + fish oil; vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3 placebo
  Arms: vitamin D placebo + fish oil; vitamin D placebo + fish oil placebo
Dietary Supplement: fish oil placebo
  Arms: vitamin D + fish oil placebo; vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine whether vitamin D or omega-3 fatty acids affect risk of infection and plasma hCAP18 levels.

ELIGIBILITY:
Participants in VITAL (NCT 01169259) are eligible to participate in this ancillary study. Please see NCT 01169259 for lists of inclusion and exclusion criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25874 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
upper respiratory infection | one year
hCAP-18 | one year

SECONDARY OUTCOMES:
lower respiratory infection | 5 years
urinary tract infection | 5 years
cellulitis | 5 years
antimicrobial-treated infection | 5 years
infection-related hospitalizations | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Manson JE, Bassuk SS, Lee IM, Cook NR, Albert MA, Gordon D, Zaharris E, Macfadyen JG, Danielson E, Lin J, Zhang SM, Buring JE. The VITamin D and OmegA-3 TriaL (VITAL): rationale and design of a large randomized controlled trial of vitamin D and marine omega-3 fatty acid supplements for the primary prevention of cancer and cardiovascular disease. Contemp Clin Trials. 2012 Jan;33(1):159-71. doi: 10.1016/j.cct.2011.09.009. Epub 2011 Oct 2. PMID 21986389
- [Background] Bassuk SS, Manson JE, Lee IM, Cook NR, Christen WG, Bubes VY, Gordon DS, Copeland T, Friedenberg G, D'Agostino DM, Ridge CY, MacFadyen JG, Kalan K, Buring JE. Baseline characteristics of participants in the VITamin D and OmegA-3 TriaL (VITAL). Contemp Clin Trials. 2016 Mar;47:235-43. doi: 10.1016/j.cct.2015.12.022. Epub 2016 Jan 6. PMID 26767629
- See also: VITAL study website — http://www.vitalstudy.org/